CLINICAL TRIAL: NCT05733026
Title: Effect of Genetic and Epigenetic Factors on the Clinical Response and Toxicity to Doxorubicin Among Egyptian Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Neven Sarhan, Lecturer, Misr International University
Other Study IDs: BC-Genetics
Record Dates: First submitted 2023-01-27; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Doxorubcin; Breast cancer; Cardiotoxicity; Gene polymorphism
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1: Breast cancer patients who developed cardiotoxic side effects in response to Doxorubicin treatment
- 2: Breast cancer patients who did not develope cardiotoxic side effects in response to Doxorubicin treatment

SUMMARY:
Recent advances in technologies, such as microarray and high-throughput sequencing, represented a deeper understanding of molecular biology, especially noncoding RNA (ncRNA). It was found that there are only <2 % of the total genome sequence as protein-coding genes while at least 98 % of the genome are transcribed into ncRNA. In the past, non-protein-coding RNAs were known as "transcription noise," but now it is obvious that ncRNAs play a crucial regulatory role in cell differentiation and organism growth and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic and localized breast cancer patients treated with Doxorubicin among chemotherapeutic protocol.
* Measurable disease.
* Age of 18 years to 80 years.
* The women of childbearing age must use an effective contraception for the duration of the study.

Exclusion Criteria:

* Breast cancer patients who had undergone radiotherapy or chemotherapy.
* Pregnant and lactating females.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to chemotherapeutic agents used.
* Any other medical or psychiatric condition or severe or chronic laboratory abnormality making the inclusion of the patient in the study inappropriate in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic and localized breast cancer patients treated with Doxorubicin
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Cardiotoxicity | 6 months
  Occurrence of dilated cardiomyopathy

SECONDARY OUTCOMES:
Nephrotoxicity | 6 months
  Occurrence of nephrotoxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided